CLINICAL TRIAL: NCT02402010
Title: Pilot Study of Adjunctive Yoga for Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Butler Hospital (Other)
Responsible Party: Principal Investigator, Lauren M. Weinstock, PhD, Associate Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB1401-001
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjunctive Yoga (Experimental): Participants may be randomized to receive up to 10 weeks of group yoga class, as an adjunct to medication treatment as usual provided by community clinicians.
  Interventions: Behavioral: Adjunctive Yoga
- Enhanced Treatment as Usual (Other): Those randomized to the Enhanced Treatment as Usual arm will follow their usual treatment plans in the community, with enhanced monitoring of symptoms and functioning through regular study assessments. With a release of information, we will provide community clinicians with a standardized report that summarizes level of symptom severity and risk, designed to aid in continuity of care.
  Interventions: Behavioral: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: Adjunctive Yoga
  Arms: Adjunctive Yoga
Behavioral: Enhanced Treatment as Usual
  Arms: Enhanced Treatment as Usual

SUMMARY:
As a practice that incorporates elements of physical exercise, controlled breathing, and meditation, yoga is gaining increasing acceptance as an adjunctive intervention for many psychiatric disorders. Although yoga has been frequently recommended as a symptom management strategy for bipolar disorder (BD), and although there is some preliminary evidence that yoga may be helpful in alleviating depressive symptoms, there are no systematic studies on the benefits - and potential risks - of the practice of yoga in BD. The primary aim of the proposed study is to develop and evaluate the feasibility, acceptability, and safety of an adjunctive yoga intervention for bipolar depression in a 10 week pilot randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Overcoming the burden of depression remains one of the most significant challenges in managing bipolar disorder. Compared to mania, depressive episodes in bipolar disorder are more frequent and considerably longer in length, with individuals spending roughly one-third to one-half of their lives suffering from depressive symptoms. Most of the difficulties with functioning at work, home, or school are due to depressive episodes, and most suicides occur in the context of a depressive (vs. manic) episode. Medication treatment of bipolar depression is not straightforward. Some individuals have a poor response to mood stabilizing medications, experience switches into mania as a result of antidepressant use, and have trouble taking their medications as prescribed. Thus, there remains a need for treatments that individuals with bipolar depression can use in addition to medication. As a practice that incorporates elements of physical exercise, controlled breathing, and meditation, hatha yoga has frequently been recommended as a way to manage bipolar disorder symptoms. There are numerous reasons why hatha yoga may be helpful for bipolar depression. First, there is some evidence that hatha yoga is useful for unipolar depression. Second, it is possible that yoga may help individuals with bipolar disorder regulate their daily routines, decrease negative depressive thoughts, and have a positive impact on biological mechanisms related to bipolar disorder. Yet to our knowledge, there have been no published studies on the benefits - and potential risks - of the practice of yoga in bipolar disorder. The primary aim of the proposed pilot study is to develop a 10 week yoga program specifically tailored to bipolar depression. We will develop an instructor manual for teaching classes and a scale for measuring instructor adherence to the manual. We will evaluate the feasibility, acceptability to patients, and safety of this program in a 10 week pilot randomized controlled trial (RCT). In this trial, we will enroll 36 participants with bipolar I/II depression, and randomly assign them to either: 1) the yoga intervention, delivered as an adjunct to treatment as usual; or 2) treatment as usual enhanced with a publicly-available bipolar disorder self-help book (ETAU). In a preliminary fashion, we will examine whether the yoga classes (compared to ETAU) appear promising in terms of reduced symptom severity and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of bipolar I or II disorder
* current major depressive episode
* at least 4 weeks of stable medication treatment as usual
* medical clearance for moderate exercise, as documented in a note from a primary care provider
* ability to understand English sufficiently well to understand consent or assessment instruments

Exclusion Criteria:

* presence of psychiatric symptoms severe enough to warrant inpatient hospitalization
* current psychotic symptoms
* active alcohol or substance use disorder
* pregnancy or plans to become pregnant within the year
* participation in more than 4 single sessions of yoga in the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology-Clinician Administered | 10 weeks

SECONDARY OUTCOMES:
Altman Self-Rating Mania Scale | 10 weeks
World Health Organization (WHO) Disability Assessment Schedule-II | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States